CLINICAL TRIAL: NCT02613910
Title: OPV117059: A Long-Term Extension Study of Ofatumumab Injection for Subcutaneous Use in Subjects With Pemphigus Vulgaris
Brief Title: Long-Term Extension Study of Ofatumumab in Subjects With Pemphigus Vulgaris
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Novartis has acquired the rights to ofatumumab and terminated the OPV116910 and OPV117059 studies. This decision is not linked to any safety consideration.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117059
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-04

CONDITIONS: Pemphigus
Keywords: Ofatumumab; Pemphigus Vulgaris; Long-Term Extension Study
MeSH Terms: conditions — Pemphigus | interventions — ofatumumab; Acetaminophen; Histamine Antagonists; Cetirizine; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ofatumumab (Experimental): t the Baseline (Bln) and wk 4 visits, Subjects will receive 40mg ofatumumab sc (Oft) (as two 20mg sc inj) and as 1 Oft 20mg sc inj every 4 wks from wk 8 through wk 56. Subjects will return to clinic 4 wks after the last dose for a follow-up (f/u) visit (wk 60). Antihistamine 10 mg and Acetaminophen/paracetamol (A/P) 1 grams(g) will be given 1-2 hours(h) before and 4 h after each dose of Oft. A/P 1 g will be supplied for self administration if needed. Prednisone/Prednisolone dose will continue to be tapered during core study period (CSP) by 1 dose level every 2 wks to <= 10 mg/day from Bln through wk 60. Upon completion of the CSP, subjects will enter Individualized f/u Period, where subjects will monitored every 12 wks for a minimum of 1 yr and for up to 2 yr, until CD19+ B-LC or IgG recover to lower limit of normal (LLN) or to the subject's Bln value from Study OPV116910 (if <LLN) or if study withdrawal criteria are met or for a maximum of 2 yr after the last dose of Oft.
  Interventions: Drug: Ofatumumab; Drug: Acetaminophen/paracetamol; Drug: Antihistamine (cetirizine or equivalent); Drug: Prednisone/Prednisolone

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab (human monoclonal antibody) will be provided as a liquid concentrate in a prefilled glass syringe with staked needle, stopper, and plunger containing 0.4 millilitre (mL) (20 mg) drug product of 50 mg/mL concentration
Drug: Acetaminophen/paracetamol — Acetaminophen/paracetamol will be supplied by study centre as 1 gram tablet, caplet, capsule or liquid for oral administration
Drug: Antihistamine (cetirizine or equivalent) — Antihistamine (cetirizine or equivalent) will be supplied by study center as 10 mg tablet, caplet, capsule or liquid for oral administration
Drug: Prednisone/Prednisolone — Prednisone/Prednisolone will be supplied from the dose range 2.5, 5, 7.5, 10, 12.5, 15, 17.5, 20, 25, 30, 40, 50, 60, 80, 100, 120, 140, 160, 180, 200, 220 and 240 mg for oral administration

SUMMARY:
This study is designed as a multi-country, multicenter, open label extension to Phase III trial OPV116910. The primary objective is to provide continued treatment with ofatumumab subcutaneous (SC) for eligible subjects who complete the OPV116910 trial in order to obtain further long term safety and tolerability information in subjects with pemphigus vulgaris receiving ofatumumab SC every 4 weeks (wk).

ELIGIBILITY:
Inclusion Criteria:

* Adult with clinically documented diagnosis of PV.
* Completed Study OPV116910 through Week 60 with one of the following outcomes:

Did not achieve remission by Week 60 of OPV116910. Achieved remission on a steroid dose >10 milligrams/day. Achieved remission on minimal steroid therapy, but is experiencing a disease flare/relapse while participating in the first year (yr)of the OPV116910 Individualized Follow up Period (It is recommended subjects are transitioned to the extension study before the steroid dose is increased).

* A woman is eligible to enter the study if she:

Is of non-childbearing potential: documented as surgically sterile (bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion) or is postmenopausal without menses for >2 years. Women who are <2 years postmenopausal are required to have menopausal status confirmed by follicle-stimulating hormone (FSH) and estradiol levels at the baseline evaluation. If FSH and estradiol levels do not provide confirmation of menopause, subject will be considered to be of childbearing potential.

Is of childbearing potential, with a negative pregnancy test at baseline, and agrees to the consistent and correct use of acceptable methods of contraception (Highly-Effective Methods for Avoiding Pregnancy) during heterosexual intercourse, beginning when the subject provides informed consent and lasting until 12 months after last dose of ofatumumab SC.

Exclusion Criteria:

* Past or current history of hypersensitivity to components of the investigational product or medically-significant adverse effects (including allergic reactions) from cetirizine (or antihistamine equivalent) or paracetamol/acetaminophen.
* Prior treatment with any of the following within the specified periods:

Medication and Other Treatment Restrictions Prior to OPV117059 Baseline Any time- Ofatumumab (Intravenous), total body irradiation, bone marrow transplantation, anti CD4; 6 weeks -Live vaccine 8 weeks- Immunosuppressive or immunomodulatory agents, including: azathioprine, cyclosporine, dapsone, mycophenolate, methotrexate, tacrolimus 6 months- Cyclophosphamide, cladribine, plasmapheresis, immunoabsorption, or immunoglobulin therapy, alemtuzumab, mitoxantrone 18 months -Rituximab or other anti CD20 treatments

* Confirmed PML or neurological findings potentially consistent with PML.
* Evidence or history of clinically significant infection or medical condition including:

Chronic or ongoing active infectious disease requiring long term systemic treatment, including, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, or active hepatitis C.

Positive test for hepatitis B surface antigen (HbsAg). For HbsAg negative, but hepatitis B core antibody positive (anti-HBc) (regardless of hepatitis B surface antibody [HbsAb] status), a hepatitis B virus deoxyribonucleic acid (HBV DNA) test will be performed and the subject will be excluded if results are positive. Consult with a physician experienced in the care and management of subjects with hepatitis B to manage/treat subjects who are anti HBc positive. Subjects who are anti-HBc positive and HBV DNA negative will continue to be monitored throughout the study.

History of positive serology for human immunodeficiency virus. Previous serious opportunistic or atypical infections. Prior history, or suspicion, of tuberculosis. A radiograph of the chest taken within 3 months before the first administration of investigational product suggests no evidence indicating current active tuberculosis or previous tuberculosis.

* Past or current malignancy, except for: Cervical carcinoma Stage 1B or less; Noninvasive basal cell and squamous cell skin carcinoma; Cancer diagnoses with a duration of complete response (remission) >5 years.
* Clinical chemistry and/or hematology laboratory values of clinical concern, in the investigator's opinion.

For subjects transitioning directly from the OPV116910 study, review central chemistry and hematology laboratory reports from the Week 48 through Week 56 visits of OPV116910.

For subjects transitioning from the Individualized Follow-up Period of OPV116910, review central chemistry and hematology laboratory reports from the most recent OPV116910 Individualized Follow-up visit. If the date of that laboratory report is more than 12 weeks from the extension study Screening visit, then the laboratory assessments need to be repeated.

For subjects with neutropenia (absolute neutrophil count <1 Giga units per liter, the neutropenia must resolve before the first dose of ofatumumab, which should occur within 4 weeks of the screening assessments.

* Electrocardiogram (ECG) showing a clinically significant abnormality or showing a Corrected QT Interval (QTc) interval >=450 millisecond (msec) (>=480 msec for subjects with bundle branch block) (ECG will be obtained during Week 60 visit of OPV116910; Repeat ECG if more than 12 weeks have elapsed).
* Significant concurrent, uncontrolled medical condition that could affect the subject's safety, impair the subject's reliable participation in the study, impair the evaluation of endpoints, or necessitate the use of medication not allowed by the protocol.
* In the Investigator's opinion, there is a reason why the subject would not be eligible for this study (eg, the subject is unable to comply with the visit schedule).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a multicounty, multicenter, open-label extension study to assess the long-term efficacy and safety of ofatumumab subcutaneous (SC) injection in participants with pemphigus vulgaris (PV), who completed the core study period of study OPV116910.
Pre-assignment Details: The study consisted of a screening visit, followed by a 56-week treatment period, a 4-week follow-up visit and a minimum of 1 year (up to 2 years) of individualized follow-up. Only 1 participant was enrolled into the study due to study termination.
Groups:
- Ofatumumab: At Baseline and Week 4 visits, participants were planned to receive 40 milligrams (mg) ofatumumab SC (2 X 20 mg); and 20 mg ofatumumab SC injections every 4 weeks from Week 8 through Week 56. Participants planned to return to clinic 4 weeks after the last dose for a Follow-up visit (Week 60). Antihistamine 10 mg and acetaminophen/paracetamol 1 grams (g) would be given 1-2 hours before and 4 hour after each dose of ofatumumab SC injection. Acetaminophen/paracetamol 1 g were to be self administered. Prednisone/prednisolone dose were to be tapered during core study period by 1 dose level every 2 weeks to <= 10 mg/day from Baseline through Week 60. Upon completion of the core study period, participants were to enter individualized Follow-up period, where participants were to be monitored every 12 weeks for a minimum of 1 year and up to 2 years.
Period: Overall Study
Arm/Group | Ofatumumab
Started | 1
Completed | 0
Not Completed | 1
Not completed — Termination of study | 1

BASELINE CHARACTERISTICS:
Population: Ofatumumab
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | NA (NA) — Age of the one participant enrolled in this study is not provided in order to ensure protection of participant identity.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Gender of the one participant enrolled in this study is not provided in order to ensure protection of participant identity.
  Male | NA — Gender of the one participant enrolled in this study is not provided in order to ensure protection of participant identity.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events(AEs) and AEs Leading to Permanent Discontinuation of Ofatumumab SC (AELD)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with AEs and those with AEs leading to permanent discontinuation of ofatumumab SC (AELD) were to be summarized. Safety Population consists of all participants enrolled in the study. No safety events were reported for the one participant enrolled.
Time Frame: Up to Week 60
Population: Safety Population. No safety events were reported for the one participant enrolled.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: Number of Participants With Severe Adverse Events
Description: Severity is a category utilized for rating the intensity of an adverse event. Participants with severe AEs were to be summarized. No serious adverse events (SAEs) were reported for the one participant enrolled.
Time Frame: Up to Week 60
Population: Safety Population. No safety events were reported for the one participant enrolled.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

3. Primary Outcome: Number of Participants With Adverse Events Related to Ofatumumab SC
Description: Participants with AEs related to ofatumumab were to be summarized. No adverse events related to ofatumumab were reported for the one participant enrolled.
Time Frame: Up to Week 60
Population: Safety Population. No adverse events related to ofatumumab were reported for the one participant enrolled.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and AEs of Special Interest (AESI)
Description: Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention, events associated with liver injury and impaired liver function were to be categorized as SAE. AEs of special interest included any opportunistic infections, serious post injection systemic reactions, progressive multifocal leukoencephalopathy (PML), hepatitis B virus infection or reactivation, severe mucocutaneous reactions (e.g., toxic epidermal necrolysis and stevens-johnson syndrome), cytopenias and cardiovascular events. Participants with SAEs and AESI were to be summarized. No serious adverse events (SAEs) or adverse events of special interest (AESI) reported.
Time Frame: Up to Week 156
Population: Safety Population. One participant was enrolled into the study and was withdrawn early due to study termination. No SAEs or AESIs were reported for this participant.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants
  Any SAE | 0
  Any AESI | 0

5. Primary Outcome: Number of Participants Withdrawn Due to Treatment-related AEs
Description: Participants withdrawn due to treatment related AEs were to be summarized. One participant was enrolled into the study and was withdrawn early due to study termination. The participant was not withdrawn due to treatment-related AEs.
Time Frame: Up to Week 60
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

6. Primary Outcome: Number of Participants With Infections
Description: All infections were planned to be monitored closely throughout the study and participants with infections were to be summarized. No cases of infection were reported for the one participant.
Time Frame: Up to Week 60
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

7. Primary Outcome: Number of Participants With Post-injection Systemic Reactions
Description: All serious post-injection systemic reactions were planned to be monitored closely throughout the study and number of participants with post-injection systemic reactions was to be summarized. No cases of post-injection systemic reactions were reported for the one participant.
Time Frame: Up to Week 60
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

8. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Number of participants with injection site reactions were planned to be summarized. No cases of injection site reaction were reported for the one participant.
Time Frame: Up to Week 60
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

9. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points
Description: SBP and DBP were to be taken at pre-dose and 4 hour post-dose on Week 4; pre-dose and 1 hour post-dose from Week 6 to Week 56; and at Follow-up visit (Week 60). Measurements were to be obtained after at least 5 minutes of rest. Baseline was to be considered as the measurement obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline value from the individual post-randomization values. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Baseline (Week 0) and up to Week 60
Population: Safety Population
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

10. Primary Outcome: Change From Baseline in Heart Rate at the Indicated Time Points
Description: Heart rate was to be taken at pre-dose and 4 hour post-dose on Week 4; pre-dose and 1 hour post-dose from Week 6 to Week 56; and at Follow-up visit (Week 60). Measurements were to be obtained in the sitting position and at the time of the blood pressure measurement. Baseline was to be considered as the measurement obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline value from the individual post-randomization values. Due to the termination of this study, analysis of this information was not performed
Time Frame: Baseline (Week 0) and up to Week 60
Population: Safety Population.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

11. Primary Outcome: Change From Baseline in Body Temperature at the Indicated Time Points
Description: Body temperature was planned to be taken at pre-dose and 4 hour post-dose on Week 4; pre-dose and 1 hour post-dose from Week 6 to Week 56; and at Follow-up visit (Week 60). Baseline was to be considered as the measurement obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline value from the individual post-randomization values. Due to termination of study, analysis of this information was not performed.
Time Frame: Baseline (Week 0) and up to Week 60
Population: Safety Population.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

12. Primary Outcome: Number of Participants With Vital Signs of Clinical Concern
Description: Participants with vitals signs of clinical concern were planned to be summarized. No vital signs of clinical concerns were present for the one participant.
Time Frame: Up to Week 60
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

13. Primary Outcome: Number of Participants With Clinically-significant Electrocardiogram (ECG) Abnormalities
Description: 12-lead ECG was planned to be taken on Baseline (Week 0) and at Follow-up visit (Week 60). No clinically significant ECG abnormalities were noted for the one participant.
Time Frame: Up to Week 60
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

14. Primary Outcome: Change From Baseline in Hemoglobin at the Indicated Time Points
Description: Blood samples were planned to be collected at Baseline (Week 0) and at Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56 and at Follow-up visit (Week 60); and at individualized Follow-up visits at Week 72, 84, 96, 108, 120, 132, 144 and 156. Baseline was to be considered as the value obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline value from the individual post-randomization values. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

15. Primary Outcome: Change From Baseline in Hematocrit at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

16. Primary Outcome: Change From Baseline in White Blood Cell (WBC) Count, Neutrophil, Lymphocyte, Basophil, Eosinophil, Monocyte, Platelet Count, Bands, Cluster of Differentiation (CD)19+ B-lymphocyte Counts, CD3, CD4 and CD8 at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

17. Primary Outcome: Change From Baseline in CD4: CD8 Ratio at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

18. Primary Outcome: Change From Baseline in Red Blood Cell (RBC) Count and Nucleated RBCs at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

19. Primary Outcome: Change From Baseline in Total Protein and Albumin at the Indicated Time Points
Description: Blood samples were planned to be collected at Baseline (Week 0) and at Week 8, 20, 28, 36, 44, 52 and at Follow-up visit (Week 60); and at individualized Follow-up visits at Week 72, 84, 96, 108, 120, 132, 144 and 156. Baseline was to be considered as the value obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline value from the individual post-randomization values. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

20. Primary Outcome: Change From Baseline in Total Bilirubin and Creatinine at the Indicated Time Points
Description: as for outcome 19
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

21. Primary Outcome: Change From Baseline in Alanine Aminotransferase, Aspartate Aminotransferase, Alkaline Phosphatase and Gamma Glutamyl Transferase at the Indicated Time Points
Description: as for outcome 19
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

22. Primary Outcome: Change From Baseline in Sodium, Potassium, Chloride, Calcium, Glucose, Bicarbonate and Blood Urea Nitrogen at the Indicated Time Points
Description: as for outcome 19
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

23. Primary Outcome: Change From Baseline in Creatinine Clearance (Calculated) at the Indicated Time Points
Description: Blood samples were plannedto be collected at Baseline (Week 0) and at Week 8, 20, 28, 36, 44, 52 and at Follow-up visit (Week 60); and at individualized Follow-up visits at Week 72, 84, 96, 108, 120, 132, 144 and 156. Baseline was to be considered as the value obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline value from the individual post-randomization values. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

24. Primary Outcome: Number of Participants With Change in Urinalysis Results
Description: Urine samples were planned to be collected at Baseline (Week 0) and at Week 8, 20, 28, 36, 44, 52 and at Follow-up visit (Week 60) for evaluation of appearance, protein, glucose, leukocyte esterase, ketones, hemoglobin, microalbumin, creatinine, microalbumin:creatinine ratio and microscopy which included RBC/high powered field, WBC/ hight powered field, epithelial cells, trichomonas, bacteria, yeast, crystals, ammonium urates, mucous threads, amorphous sediment and casts. Baseline was to be considered as the measurement obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline from the individual post-randomization measurements. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

25. Primary Outcome: Change From Baseline in Urine Power of Hydrogen (pH) at the Indicated Time Points
Description: Urine samples were plannedto be collected at Baseline (Week 0) and at Week 8, 20, 28, 36, 44, 52 and at Follow-up visit (Week 60) for evaluation of pH. Baseline was to be considered as the measurement obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline from the individual post-randomization measurements. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

26. Primary Outcome: Change From Baseline in Specific Gravity of Urine
Description: Urine samples were planned to be collected at Baseline (Week 0) and at Week 8, 20, 28, 36, 44, 52 and at Follow-up visit (Week 60) for evaluation of urine specific gravity. Baseline was to be considered as the measurement obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline from the individual post-randomization measurements. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

27. Primary Outcome: Number of Participants With Laboratory Results of Potential Clinical Concern
Description: Blood samples were planned to be collected at Baseline (Week 0) and at Week 8, 20, 28, 36, 44, 52 and at Follow-up visit (Week 60); and at individualized Follow-up visits at Week 72, 84, 96, 108, 120, 132, 144 and 156 for evaluation of clinical chemistry parameters; and at Baseline (Week 0) and at Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56 and at Follow-up visit (Week 60); and at individualized Follow-up visits at Week 72, 84, 96, 108, 120, 132, 144 and 156 for evaluation of hematology parameters. No laboratory values of potential clinical concern were identified for this one participant.
Time Frame: Up to Week 156
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 1
Participants | 0

28. Primary Outcome: Change From Baseline in Immunoglobulin (Ig) A, IgM, and IgG Levels
Description: Blood samples for IgA, IgM, and IgG analysis were planned to be collected at Baseline (Week 0) and at Week 12, 24, 36, 48 and at Follow-up visit (Week 60); and at individualized Follow-up visits at Week 72, 84, 96, 108, 120, 132, 144 and 156. Baseline was to be considered as the value obtained on Week 0. The change from Baseline was to be calculated by subtracting the Baseline value from the individual post-randomization values. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

29. Secondary Outcome: Time to Sustained Remission on Minimal Steroid Therapy
Description: Time to sustained remission on minimal steroid therapy is the time from Baseline (Week 0) to the time the participant initially tapered his/her oral prednisone/prednisolone dose to <=10 mg/day and maintained <=10 mg/day of oral prednisone/prednisolone with no new or non-healing (established) lesions for >= 8 weeks and maintained that status until Week 60. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

30. Secondary Outcome: Duration of Remission on Minimal Steroid Therapy
Description: Duration of remission on minimal steroid therapy is the total time (sum) of all periods of remission while on minimal steroid therapy (oral prednisone/prednisolone dose <=10 mg/day) up to Week 60. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

31. Secondary Outcome: Number of Participants Achieving Sustained Remission on Minimal Steroid Therapy by Week 60
Description: Sustained remission on minimal steroid therapy is the time from Baseline (Week 0) to the time the participant initially tapered his/her oral prednisone/prednisolone dose to <=10 mg/day and maintained <=10 mg/day of oral prednisone/prednisolone with no new or non-healing (established) lesions for >=8 weeks and maintained that status until Week 60. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

32. Secondary Outcome: Time to Remission Off Steroid Therapy by Week 60
Description: Remission is the absence of new or non-healing (established) lesions for >=8 weeks. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

33. Secondary Outcome: Number of Participants Achieving Remission While Off Steroid Therapy by Week 60
Description: as for outcome 32
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

34. Secondary Outcome: Number of Participants Achieving Remission on Minimal Steroid Therapy
Description: Remission is defined as absence of new or non-healing (established) lesions for >=8 weeks and minimal steroid therapy is defined as an oral prednisone/prednisolone dose of <=10 mg/day. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

35. Secondary Outcome: Time to Remission on Minimal Steroid Therapy
Description: Time to remission on minimal steroid therapy is the time from Baseline to the time the participant initially tapered his/her oral prednisone/prednisolone dose to <=10 mg/day and maintained <=10 mg/day of oral prednisone/prednisolone with no new or non-healing (established) lesions for >=8 weeks by Week 60. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

36. Secondary Outcome: Duration of Remission After Completing the Ofatumumab SC Treatment Course
Description: Duration of remission after completing the ofatumumab SC treatment course was to be assessed during the individualized Follow-up period for participants who were in remission on minimal steroid therapy by Week 60. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

37. Secondary Outcome: Time to Initial Flare/Relapse by Week 60
Description: Time to initial flare/relapse is time from Baseline to the time of appearance of >= 3 new lesions within 1 month that do not heal spontaneously within 1 week, or to the time when there is an extension of lesions that were present at the Baseline visit. The appearance of 1 or 2 new lesions was not to be considered a flare/relapse. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

38. Secondary Outcome: Number of Participants Who do Not Flare/Relapse
Description: It was planned to assess participants with out an appearance of >= 3 new lesions within 1 month that do not heal spontaneously within 1 week, or an extension (worsening) of lesions that were present at the Baseline visit. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

39. Secondary Outcome: Number of Participants Who do Not Flare/Relapse on Minimal Steroid Therapy
Description: It was planned to assess as participants who achieved remission on minimal steroid therapy and did not subsequently have a flare/relapse of disease by Week 60. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

40. Secondary Outcome: Time to Initial Flare/Relapse After Completing the Ofatumumab SC Treatment Course
Description: It is the time from Baseline to the time of appearance of >=3 new lesions within 1 month that do not heal spontaneously within 1 week, or to the time when there is an extension of lesions that were present at the Baseline visit. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

41. Secondary Outcome: Time to Initial Flare/Relapse After Completing the Ofatumumab SC Treatment Course During the Individualized Follow-up Period
Description: as for outcome 40
Time Frame: Up to Week 156
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

42. Secondary Outcome: Number of Days Minimal Steroid Therapy is Maintained by Week 60
Description: Minimal steroid therapy is an oral prednisone/prednisolone dose of <= 10 mg/day. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

43. Secondary Outcome: Number of Days a Participant is Off Steroid Therapy by Week 60
Description: Number of days, a participant did not require steroid therapy was observed and summarized. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

44. Secondary Outcome: Cumulative Dose of Corticosteroids
Description: Cumulative dose of corticosteroids was calculated to evaluate steroid exposure and reductions in steroid dose while maintaining disease control. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 60
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

45. Secondary Outcome: Number of Participants With Positive Human Anti-human Antibody (HAHA) Immune Response
Description: Blood samples for HAHA titer analysis were planned to be collected at Baseline (Week 0) and at Week 12, 24, 36, 48 and at Follow-up visit (Week 60); and at individualized Follow-up visit at Week 72. Due to the termination of this study, analysis of this information was not performed.
Time Frame: Up to Week 72
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

46. Secondary Outcome: Titer of Human Anti-human Antibody
Description: as for outcome 45
Time Frame: Up to Week 72
Population: Safety Population. Due to the termination of this study, 0 participants were analyzed.
Arm/Group | Ofatumumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: On-treatment non-serious AEs were to be collected from the start of the study treatment up to Week 60 and SAEs were to be collected from start of the study up to Week 156. No on-treatment non-serious AEs were reported for the one participant.
Description: On treatment SAEs and non-serious AEs were to be reported for the Safety Population. No on-treatment non-serious AEs were reported for the one participant.
Arm/Group | Ofatumumab
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.